CLINICAL TRIAL: NCT04118426
Title: Cognitive Function After Radiation Therapy for Brain Tumours
Acronym: WP-12-pre
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Morten Høyer, Professor, University of Aarhus
Other Study IDs: WP-12's precursor
Record Dates: First submitted 2018-06-01; First posted 2019-10-08 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Primary Brain Tumor; Radiation Toxicity
Keywords: Cognitive function
MeSH Terms: conditions — Brain Neoplasms; Radiation Injuries | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Radiotherapy group: Patients receiving radiotherapy after surgery for brain tumor
  Interventions: Radiation: Cognitive testing
- No radiotherapy group: Patients NOT receiving radiotherapy after surgery for brain tumor
  Interventions: Radiation: Cognitive testing

INTERVENTIONS:
Radiation: Cognitive testing — Patients will have their cognitive function tested by the use of standardized cognitive test and fill in questionnaires.
  Cognitive function will be assessed by standardized cognitive tests: Hopkins verbal learning test (HVLT), Trail Making Test part A and B (TMT A and TMT B), Pased Auditory Test (PASAT), Wechsler Adult Intelligence Scale coding and digit span (WAIS-IV), Controlled Oral Word Association Test (Cowat) and STROOP colour and word test (STROOP)
  Questionnaire include; Quality of life; EORTC QlQ-C30 (QlQ-C30), FACIT-Fatigue Scale (Version 4) (FACIT), Pittsburg Sleep Quality Index (PSQI), Hospital Anxiety and Depression Scale (HADS), Patient's Assessment of Own Functioning Inventory (PAOFI).

SUMMARY:
This study will assess cognitive function in adult patients with a primary brain tumour treated with surgical resection with or without radiation therapy (RT). All types of brain tumours apart from glioblastoma will be included

DETAILED DESCRIPTION:
RT to brain tumours causes cognitive dysfunction. The extent of RT induced changes in cognitive function and radio-sensitivity of the brain is unknown. RT with protons instead of photons spares the healthy brain tissue more and is believed to reduce the risk of cognitive dysfunction. There is modest knowledge on which parts of the brain the investigators need to spare, to prevent cognitive dysfunction.

The study is a cross sectional study assessing cognitive function in patients with brain tumours previously treated with RT compared to a similar non irradiated group. 104 patients with specified brain tumours from Aarhus University Hospital treated in the period 2006-2016 will be included. The patients will do patient reported outcome (PRO) and undergo neuropsychological assessment with standardized tests: They will do this prior to RT treatment and ½, 1, 3 and 5 years afterwards. The PRO's included measures on quality of life, fatigue, sleep, depression, anxiety, and socio demografica. The standardized tests are: Trail making Test (TMT); Hopkins Verbal Learning Test (HVLT); Controlled Oral Word Association Test (COWAT) - Animals and S; Coding and Digit Span from WAIS-IV; Paced Auditory Serial Addition Test (PASAT). The correlation between cognitive scores and RT dose-volume parameters to specific areas in the brain will be tested.

ELIGIBILITY:
Inclusion Criteria:

* The participant must be 18 years or older and Danish speaking.
* Performance status 0-2
* Capable of cooperating on testing
* Diagnosed with one of the following diagnoses according to WHO 2016 classification 16 and been treated between 2006 and 2016

  1. ZM93803 glioma (exclusive glioblastoma)
  2. ZM9401/3 anaplastic astrocytoma, IDH mutant
  3. ZM9400/3 diffuse astrocytoma, IDH-mutant
  4. ZM9411/3 gemistocytisk astrocytoma, IDH mutant
  5. ZM9400/3 diffuse astrocytoma, NOS
  6. ZM9451/3 anaplastic oligodendroglioma, IDH mutant and 1p/19q-co deleted
  7. ZM9450/3 oligodendroglioma, IDH mutant and 1p/19q-co deleted
  8. ZM9450/3 oligodendroglioma, NOS
  9. ZM9451/3 anaplastic oligodendroglioma, NOS
  10. ZM9530/0 meningioma
  11. ZM9470/3 medulloblastoma, NOS
  12. DD352A pituitary adenoma
  13. Other rare brain tumours including skull base sarcomas

      -

      Exclusion Criteria:

      Performance status 3-4 Progression after radiation therapy

      -

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with a primary brain tumour grade I-III
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2018-02-02 (Actual); Study Completion 2018-04-12 (Actual)

PRIMARY OUTCOMES:
Memory impairment (as assessed by the HVLT-r) | 1-10 years after treatment
  To examine the correlation between memory impairment (assessed by HVLT-r) and mean dose to the hippocampus.
Neurocognitive function | 1-10 years after treatment
  Examine correlations cognitive decline and subvolumes of the brain. Cognitive function will be assessed by standardized cognitive tests: Hopkins verbal learning test (HVLT), Trail Making Test part A and B (TMT A and TMT B), Pased Auditory Test (PASAT), Wechsler Adult Intelligence Scale coding and digit span (WAIS-IV), Controlled Oral Word Association Test (Cowat) and STROOP colour and word test (STROOP). Measures on cognitive test is time in seconds or number of "corrects".

SECONDARY OUTCOMES:
Global Health - Quality of life | 1-10 years after treatment
  Assessed by questionnaire; EORTC QlQ-C30 in order to examine the level of quality of life in brain tumour patients who has received radiation therapy
Fatigue | 1-10 years after treatment
  Assessed by questionnaire: FACIT-Fatigue scale (version 4) in order to explore the level of fatigue in brain tumour patients who has received radiation therapy
Sleep quality | 1-10 years after treatment
  Assessed by questionnaire:Pittsburg Sleep Quality INDEX, PSQI in order to explore the level of quality of sleep in brain tumour patients who has received radiation therapy
Depression/Anxiety | 1-10 years after treatment
  Assessed by questionnaire: Hospital anxiety and depression Scale (HADS) in order to explore level of depression and anxiety in patients treated with radiation therapy for their brain tumour
Patients assessment of own cognitive function | 1-10 years after treatment
  Assessed by questionnaire; Patient's Assessment of Own Functioning Inventory (PAOFI), in order to assess patients own perception of cognitive function

CONTACTS AND LOCATIONS:
Overall Officials: Morten Høyer, M.D., Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Region Midt, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haldbo-Classen L, Amidi A, Lukacova S, Wu LM, Oettingen GV, Lassen-Ramshad Y, Zachariae R, Kallehauge JF, Hoyer M. Cognitive impairment following radiation to hippocampus and other brain structures in adults with primary brain tumours. Radiother Oncol. 2020 Jul;148:1-7. doi: 10.1016/j.radonc.2020.03.023. Epub 2020 Mar 28. PMID 32298906